CLINICAL TRIAL: NCT03055572
Title: Olfactory Training for Olfactory Dysfunction in Chronic Rhinosinusitis
Brief Title: Olfactory Training in Chronic Rhinosinusitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Staffing issues resulted in the closure of the study prior to any participants being enrolled.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Thomas S. Edwards, MD, Medical House Staff, Department of Otolaryngology - Head and Neck Surgery, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00094289
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Olfactory Dysfunction
Keywords: Rhinitis; Chronic Rhinosinusitis; Olfactory Training
MeSH Terms: conditions — Rhinitis | interventions — Olfactory Training; Oils, Volatile

STUDY DESIGN:
Intervention Model Description: Participants are randomized into one of three study arms: essential oil arm, pure fragrance oil arm, and control arm.
Who Masked: Participant
Masking Description: Participants assigned to the either of the olfactory training arms will not know if they are in the essential oil arm or the pure fragrance oil arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Olfactory Training with Essential Oils (Experimental): Participants assigned to this group will do olfactory training using essential oils, while continuing the medical therapy prescribed by their provider.
  Interventions: Other: Olfactory Training with Essential Oils
- Olfactory Training with Pure Fragrance Oils (Active Comparator): Participants assigned to this group will do olfactory training using pure fragrance oils, while continuing the medical therapy prescribed by their provider.
  Interventions: Other: Olfactory Training with Pure Fragrance Oils
- Control Group (No Intervention): The control group will continue the medical therapy prescribed by their provider.

INTERVENTIONS:
Other: Olfactory Training with Essential Oils — Participants will be instructed to sniff one of four provided odors for approximately 10 seconds followed by a 10 second break before repeating with each successive odor for a total of 5 minutes. Essential oils will be used for the odors. The intervention will be completed in the morning before breakfast and in the evening before bed. Participants will document compliance by completing a log of olfactory training sessions.
  Arms: Olfactory Training with Essential Oils
Other: Olfactory Training with Pure Fragrance Oils — Participants will be instructed to sniff one of four provided odors for approximately 10 seconds followed by a 10 second break before repeating with each successive odor for a total of 5 minutes. Pure fragrance oils will be used for the odors. The intervention will be completed in the morning before breakfast and in the evening before bed. Participants will document compliance by completing a log of olfactory training sessions.
  Arms: Olfactory Training with Pure Fragrance Oils

SUMMARY:
Persons with a loss of sense of smell, who agree to participate in this study, will be assigned to one of three groups: two groups will have smell training and the third group will not do smell training. Participants assigned to one of the smell training groups will be asked to smell four different odors in rotation for five minutes two times per day, a total of 10 minutes of participation per day, for 12 weeks. One smell training group will be given odors made of fragrance oils to use for smell training. The other smell training group will be given odors made of essential oils to use. Participants in all groups will continue taking all medications and nasal rinses for sinusitis as prescribed by their doctor.

DETAILED DESCRIPTION:
Problems with the ability to smell are referred to as olfactory dysfunction (OD). This condition is a widespread issue. 10-20% of all adults have OD, with 15 million individuals in the US self-reporting it in the past year. Chronic rhinosinusitis (CRS) is defined as 12 weeks or longer of non-clear nasal drainage, nasal congestion, facial pain or pressure, and/or decreased sense of smell. CRS is a common cause of OD. Up to 78% of patients with CRS reporting decreased sense of smell.

Several previous studies have shown a beneficial treatment option for OD called olfactory training (OT). OT consists of smelling different odors several times per day, every day for several months. These studies have shown that OT improves the sense of smell in patients who lost their sense of smell due to acute infection, head trauma, or diseases of the brain like Parkinson's disease. OT has not, however, been studied previously as a treatment for OD due to CRS.

The proposed study will use a randomized controlled trial to investigate if OT is effective for the treatment of OD in CRS. It will also investigate if widely available and lower cost odors, called essential oils, are as effective as traditionally used, pure fragrance oils, for OT in CRS. Lastly, the modified Questionnaire of Olfactory Disorders (mQOD) will be tested to determine if it can be used as a valid measure for monitoring patient's response to treatment.

Patients diagnosed with CRS who report that their sense of smell is diminished on a standard intake survey given to all patients will be recruited for the study by their treating practitioner. Once enrolled and consented, the subject will take the mQOD and then undergo a baseline Brief Smell Identification Test (BSIT) test. They will then be randomly assigned to one of three groups. The subjects in two groups (n = 50 subjects per group) will receive OT while the subjects in the third group (n = 50 subjects) will serve as a control group and will not receive OT. Subjects in the OT groups will be asked to smell four different odors in rotation for five minutes two times per day, a total of 10 minutes of participation per day. Half of the patients assigned to the OT group will be given odors made of fragrance oils. The other half will be given odors made of essential oils to use. Patients will be blinded to whether they were given fragrance oils or essential oils. Subjects in the OT groups will be asked to record each training session in a provided journal.

All subjects regardless of group will be sent an electronic version of the mQOD via email after the first and second month. Regardless of which group subjects are assigned, they will continue taking all medications and treatments for CRS as if they were not enrolled in this study. After three months, all subjects will again complete this survey as well as a second BSIT test. This study will determine if a) OT is an effective treatment for OD due to CRS, b) essential oils are as effective as pure fragrance oils for OT in CRS, and c) if the mQOD can be used to monitor treatments for OD in CRS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic rhinosinusitis (CRS) by consensus criteria from the International Consensus Statement on Allergy and Rhinology: Rhinosinusitis (ICAR:RS)
* Self-reports that decreased sense of smell/taste is moderate, severe, or as bad as it can be on the Sino-Nasal Outcome Test (SNOT)
* Trial of saline irrigations and topical nasal corticosteroids for >3 weeks

Exclusion Criteria:

* Diagnosis of cystic fibrosis, congenital anosmia, or neurocognitive disorder
* History of sinonasal tumor or anterior skull base resection
* Development of olfactory dysfunction (OD) immediately following facial trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-12-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Changes in Brief Smell Identification Test (BSIT) | Baseline, Week 12
  The Brief Smell Identification Test (BSIT) is a 12-question scratch-n-sniff test to evaluate sense of smell. Score ranges from 0 to 12. Higher BSIT score indicate a better sense of smell. BSIT scores ≥ 9 is considered normal. Lower BSIT scores (≤ 8) indicate olfactory dysfunction. A change in BSIT by 1 is considered clinically significant.
Changes in modified Questionnaire of Olfactory Disorders (mQOD) score | Baseline, Week 4, Week 8, and Week 12
  The modified Questionnaire of Olfactory Disorders (mQOD) is a 17-item survey assessing quality of life in individuals with olfactory disorder. Respondents rate how much they agree with statements about how much their daily lives, social encounters, and feelings of safety are impacted by loss of smell by selecting "I agree" , "I agree partly", "I disagree partly" or "I disagree".

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Edwards, MD, Principal Investigator — Emory University

IPD SHARING:
Plan to Share IPD: No